CLINICAL TRIAL: NCT03871049
Title: Effect of Adding Dexamethasone to Intrathecal Bupivacaine on Blood Sugar of Patients Undergoing Diabetic Foot Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman A. Ismail, assistant profesor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 01003060566
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Placebo Comparator): intathecal bupivacaine
  Interventions: Drug: Bupivacaine
- group 2 (Active Comparator): intrathecal bupivacaine with dexamethasone
  Interventions: Drug: Bupivacaine with dexamethasone

INTERVENTIONS:
Drug: Bupivacaine with dexamethasone — bupivacaine with dexamethasone
  Arms: group 2
Drug: Bupivacaine — bupivacaine
  Arms: group 1

SUMMARY:
effect of intrathecal dexamethasone on blood sugar of dietetic patients

ELIGIBILITY:
Inclusion Criteria:

* control diabetic patients will undergo foot surgeries.

Exclusion Criteria:

* The exclusion criteria included patient refusal, patients with major cardiac, respiratory, renal, hepatic disorders or uncontrolled diabetes mellitus, history of chronic use of analgesic medication or hypersensitivity to drugs under investigation, any contraindication to regional anesthesia, namely; patients with coagulopathy infection at puncture site, backache, spine deformity or prior surgery, neuromuscular disorders or psychic disturbances

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
blood sugar | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt